CLINICAL TRIAL: NCT04930146
Title: To Evaluate the Functional Recovery Effect of Bloodletting Puncture at Jing-well Points on Acute Brain Injury Patients
Brief Title: Functional Recovery Effect of Bloodletting Puncture at Jing-well Points on Acute Brain Injury Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202100683A3
Record Dates: First submitted 2021-06-09; First posted 2021-06-18 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Traumatic Brain Injury (TBI)
Keywords: Traumatic brain injury, TBI; Bloodletting; acupuncture
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Acupuncture Therapy; Bloodletting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group (Severe) (Experimental): A patient's Glasgow Coma Score (GCS) between 5-8
  1. Conventional treatment and bloodletting at the well points of both hands and feet and acupuncture in DU26, DU24 3 times per week for 4 weeks, total 12 treatments.
  2. Evaluating the meridian energy by M.E.A.D
  Interventions: Other: acupuncture and bloodletting
- Control group (Severe) (No Intervention): A patient's Glasgow Coma Score (GCS) between 5-8
  1. Conventional treatment.
  2. Evaluating the meridian energy by M.E.A.D
- Intervention group (Moderate) (Experimental): A patient's Glasgow Coma Score (GCS) between 9-13
  1. Conventional treatment and bloodletting at the well points of both hands and feet and acupuncture in DU26, DU24 3 times per week for 4 weeks, total 12 treatments.
  2. Evaluating the meridian energy by M.E.A.D
  Interventions: Other: acupuncture and bloodletting
- Control group (moderate) (No Intervention): A patient's Glasgow Coma Score (GCS) between 9-13
  1. Conventional treatment.
  2. Evaluating the meridian energy by M.E.A.D

INTERVENTIONS:
Other: acupuncture and bloodletting — bloodletting at the well points of both hands and feet and acupuncture in DU26, DU24 3 times per week for 4 weeks, total 12 treatments.
  Arms: Intervention group (Moderate); Intervention group (Severe)

SUMMARY:
Traumatic brain injury (Traumatic brain injury, TBI) can be derived from various forms of injury, including blunt trauma, penetrating or acceleration/deceleration force caused by head injury.There are some study data show that acupuncture treatment has a superficial effect on the prognosis of traumatic brain injury and can limit the progression of secondary brain injury, but the effect of early bloodletting at the Jing-points on TBI patients still unknown. In our study, the investigators have proposed a randomized, controlled study design and plan to evaluate the efficacy and safety of Jing-point puncture to improve consciousness and neurological function in patients with TBI. In addition, an objective meridian instrument analysis was added to analyze the energy distribution in the meridian of TBI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with moderate to severe head injury are admitted to the ICU (Intensive Care Unit). patient with stable vital sign and the GCS (Glasgow coma volume) between 5-13 will be included.
2. Patient with normal consciousness and no cognitive or motor function disease before brain injury.
3. Patient aged between 20 to 80 years old and is willing to sign the consent (the agent can sign on behalf of patient).

Exclusion Criteria:

1. Patients who are vital sign unstable and with severe complication.
2. Patients combined with other terminal illness such as cancer in terminal stage, liver failure, end stage renal failure and so on.
3. Pregnant patients.
4. Any other conditions deemed unsuitable by the physician in charge.
5. Patients (agent of the patient) who did not sign the consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
GCS(Glasgow Coma Scale) | 4 weeks
  To assess the recovery of consciousness. Lower GCS scores are correlated with higher risk of death.
Barthel index | 4 weeks
  To assess the activities of daily life.
Muscle power | 4 weeks
  To assess the recovery of muscle power.
mGOS(Modified Glasgow Outcome Score) | 4 weeks
  To assess the neurological outcomes, score 1 to 5. the higher the score, the better outcome.
RTS (Revised Trauma Score) | 4 weeks
  To assess the physiologic condition of patients. The Revised Trauma Score is made up of a three categories: Glasgow Coma Scale, systolic blood pressure, and respiratory rate. The score range is 0-12. A lower score indicates a higher severity of injury.

SECONDARY OUTCOMES:
Meridian energy assessment | 4 weeks
  To assess meridian energy by Meridian Energy Analysis Device (M.E.A.D. )

CONTACTS AND LOCATIONS:
Overall Officials: wei Ling Chou, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No